CLINICAL TRIAL: NCT06525298
Title: A Phase 1/2, Open Label Trial to Investigate the Safety, Tolerability, and Preliminary Efficacy of EIS-12656 as Single Agent and in Combination With a Poly-ADP Ribose Polymerase (PARP) Inhibitor or Trastuzumab Deruxtecan (T-DXd), an Antibody Drug Conjugate (ADC), in Participants With Specified Solid Tumors
Brief Title: EIS-12656 as Single Agent and in Combination in Patients With Specified Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisbach Bio GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EIS-12656C01
Record Dates: First submitted 2024-07-17; First posted 2024-07-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Advanced Solid Tumor; Homologous Recombination Deficiency; HRR Deficiency
MeSH Terms: interventions — olaparib; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- EIS-12656 Dose Escalation (Experimental)
  Interventions: Drug: EIS-12656
- Dose Expansion Module 1 (EIS-12656 Monotherapy) (Experimental)
  Interventions: Drug: EIS-12656
- Dose Expansion Module 2 (EIS-12656 + Olaparib) (Experimental): EIS-12656 will be given in combination with Olaparib
  Interventions: Drug: EIS-12656; Drug: Olaparib
- Dose Expansion Module 3 (EIS-12656 + T-DXd) (Experimental): EIS-12656 will be given in combination with Trastuzumab deruxtecan
  Interventions: Drug: EIS-12656; Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: EIS-12656 — EIS-12656 tablets given daily
Drug: Olaparib — as per USPI/SmPC
  Arms: Dose Expansion Module 2 (EIS-12656 + Olaparib)
Drug: Trastuzumab deruxtecan — as per USPI/SmPC
  Other Names: Enhertu
  Arms: Dose Expansion Module 3 (EIS-12656 + T-DXd)

SUMMARY:
This trial investigates a new drug, EIS-12656, in participants with specified advanced solid tumors carrying pre-specified mutations. The trial consists of a dose escalation part (Phase 1) and a dose expansion part (Phase 2).

DETAILED DESCRIPTION:
The trial is a Phase 1/2, open label, uncontrolled trial to investigate the safety and preliminary efficacy of EIS-12656 alone or in combination with a PARPi or T-DXd in patients with specified advanced or metastatic solid tumors with homologous recombination deficient (HRD) mutations.

In the Phase 1 dose escalation phase participants will receive ascending doses of EIS-12656 to evaluate the safety and tolerability and to determine an effective and safe dose for the Phase 2 part.

In the Phase 2 dose expansion phase participants will either receive EIS-12656 monotherapy at the recommended Phase 2 dose (RP2D) (Module 1) or EIS-12656 in combination with a PARPi or T-DXd (Modules 2 and 3). The objective is to evaluate the safety and tolerability and anti-tumor activity of EIS-12656 alone or in combination.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent locally advanced or metastatic solid tumors
* Homologous recombination deficient mutations
* Progressed on at least on prior line of treatment or intolerant to additional effective standard therapy
* Measurable disease (RECIST 1.1 Criteria)
* Adequate organ and bone marrow function
* ECOG Performance Status 0 or 1
* Life expectancy > 3 months

Exclusion Criteria:

* History or evidence of any clinically relevant gastrointestinal disease
* Radiation therapy within ≤2 weeks
* Significant cardiovascular disease
* Uncontrolled, active, symptomatic brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of participants experiencing treatment-emergent adverse events (TEAEs) | From screening until end of treatment follow-up (45 days after last dose) (up to 7 months)
  Number and percentage of participants with adverse events, serious adverse events, adverse events of special interest including changes in safety lab parameters, physical examinations, vital signs, and electrocardiogram (ECG)
Number and percentage of participants experiencing a dose limiting toxicity (DLT) (dose escalation part only) | Within 21 days of first dose
  A DLT is defined as an EIS-12656 related adverse event during the first treatment cycle that meets the criteria outlined in the study protocol

SECONDARY OUTCOMES:
Maximum plasma concentration of EIS-12656 (Cmax) | At pre-defined intervals from pre-dose Day 1 to Day 29
  The concentration of EIS-12656 in plasma will be determined (Cmax will be derived)
Area under the curve (AUC0-24) | At pre-defined intervals from pre-dose Day 1 to Day 29
  The AUC0-24 reflects the actual body exposure to drug over the last 24h dosing interval
Time to maximum concentration (Tmax) | At pre-defined intervals from pre-dose Day 1 to Day 29
  The concentration of EIS-12656 in plasma will be determined (Tmax will be derived)
Overall Response Rate | From screening to disease progression (approximately 1 year)
  Overall response rate defined as percentage of participants with the best overall response of confirmed CR or confirmed PR according to RECIST v1.1
Duration of Response | From screening to disease progression or death (approximately 1 year)
  Time from first response to progression or death, as defined by RECIST 1.1
Progression Free Survival | From screening to disease progression or death (approximately 1 year)
  Time from first dose of EIS-12656 to progression or death, as defined by RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Yap, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No